CLINICAL TRIAL: NCT00089843
Title: IGF-1 and Bone Loss in Women Anorexia Nervosa
Brief Title: Bone Loss in Women With Anorexia Nervosa
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Karen Klahr Miller, MD, Chief, Neuroendocrine Unit, Massachusetts General Hospital
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 5 R01 DK052625 (completed); R01DK052625 (NIH); 1UL1RR025758 (NIH)
Record Dates: First submitted 2004-08-16; First posted 2004-08-17 (Estimated); Results first posted 2012-06-01 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Anorexia Nervosa
Keywords: Eating Disorders; Osteopenia
MeSH Terms: conditions — Anorexia Nervosa; Feeding and Eating Disorders; Bone Diseases, Metabolic | interventions — Testosterone; Intrinsa; Risedronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 2 (Active Comparator): Placebo Actonel (risedronate) and active testosterone patch
  Interventions: Drug: Testosterone; Drug: Placebo Actonel (risedronate)
- 3 (Active Comparator): Active Actonel (risedronate) and active testosterone patch
  Interventions: Drug: Testosterone; Drug: Actonel (risedronate)
- 4 (Active Comparator): Active Actonel (risedronate) and placebo testosterone
  Interventions: Drug: Actonel (risedronate); Drug: Placebo testosterone
- 1 (Placebo Comparator): Placebo testosterone patch and placebo Actonel (risedronate)
  Interventions: Drug: Placebo Actonel (risedronate); Drug: Placebo testosterone

INTERVENTIONS:
Drug: Testosterone — Testosterone patch 150mcg daily
  Other Names: Intrinsa
  Arms: 2; 3
Drug: Actonel (risedronate) — Actonel (risedronate) 35mg PO one time weekly
  Other Names: Actonel
  Arms: 3; 4
Drug: Placebo Actonel (risedronate) — Placebo tablet identical in appearance to active Actonel (risedronate) tablet
  Arms: 1; 2
Drug: Placebo testosterone — Placebo patch identical in appearance to testosterone patch
  Arms: 1; 4

SUMMARY:
Women with Anorexia Nervosa have been found to have low bone density. The study will determine whether administration of low doses of a natural hormone, testosterone and/or risedronate, a medication to help prevent bone breakdown will improve or prevent bone loss in this condition.

DETAILED DESCRIPTION:
II. SPECIFIC AIMS

Severe osteopenia is a prevalent complication of anorexia nervosa (AN), affecting over half of all women with this disease. Loss of 25-50% of total bone mass occurs frequently and is often permanent. Although anorexia nervosa affects from 0.5-1.0% of college age women, no successful therapeutic interventions have been developed for osteoporosis in this population. Bone loss in anorexia nervosa is characterized by reduced bone formation coupled with increased bone resorption. Anorexia nervosa results in a deficiency of testosterone. Testosterone administration reduces bone resorption and data suggest that low-dose testosterone replacement therapy can increase surrogate markers of bone formation. Bisphosphonates are now well established to decrease bone resorption and improve bone density in severely osteopenic postmenopausal women. However, there are few data regarding the use of this antiresorptive therapy in women with severe pre-menopausal bone loss. Our preliminary data demonstrate that administration of a bisphosphonate decreases bone resorption and increases bone mass in women with AN after 6 and 9 months. These are the first data to demonstrate a striking increase in bone density in such women. We will test the hypothesis that a combined strategy to increase bone formation and decrease bone resorption by combining testosterone with a bisphosphonate will increase bone mass in anorexia nervosa.

The following hypotheses will be tested:

Specific Aim 1. Testosterone, a nutritionally dependent bone trophic factor, is a critical determinant of decreased bone formation in anorexia nervosa, and administration of physiologic testosterone will increase bone formation and lean body mass in this disease

We will investigate in women with anorexia nervosa whether:

A. Bone formation is reduced in association with low serum testosterone B. Testosterone deficiency is due to a combination of ovarian and adrenal defects resulting from undernutrition C. Testosterone administration reverses testosterone deficiency leading to an acute and sustained increase in bone formation and a decrease in bone resorption D. Administration of physiologic testosterone replacement stimulates increases in IGF-I levels in women with anorexia nervosa, a mechanism for increased bone formation and bone density E. Administration of physiologic testosterone replacement increases lean body mass, a major determinant of bone density

Specific Aim 2. Long-term (12 months) physiologic testosterone administration combined with a bisphosphonate increases bone density by a dual anabolic and anti-resorptive strategy

We will investigate in women with anorexia nervosa whether:

A. Physiologic testosterone administration increases bone density B. Administration of a bisphosphonate decreases the excessive state of bone resorption and increases bone density C. Co-administration of physiologic testosterone replacement and a bisphosphonate increases bone density to a greater degree than testosterone or a bisphosphonate alone by increasing bone formation and decreasing bone resorption

ELIGIBILITY:
Inclusion Criteria:

* Anorexia Nervosa,
* Over 18,
* Female,
* Decreased bone density

Exclusion Criteria:

* Medications to increase bone density

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2003-06; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Klibanski, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Miller KK, Wexler TL, Zha AM, Lawson EA, Meenaghan EM, Misra M, Binstock AB, Herzog DB, Klibanski A. Androgen deficiency: association with increased anxiety and depression symptom severity in anorexia nervosa. J Clin Psychiatry. 2007 Jun;68(6):959-65. doi: 10.4088/jcp.v68n0621. PMID 17592924

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Actonel and Active Testosterone Patch: Placebo Actonel tablet weekly and active testosterone patch (starting dose 150 mcg daily; increased to 300 mcg daily in subjects whose levels remained below the median on the initial dose)
- Active Actonel and Active Testosterone Patch: Active Actonel tablet (35 mg weekly) and Active Testosterone patch (starting dose 150 mcg daily; increased to 300 mcg daily in subjects whose levels remained below the median on the initial dose)
- Active Actonel and Placebo Testosterone: Active Actonel tablet (35 mg weekly) and Placebo Testosterone Patch
- Placebo Testosterone Patch and Placebo Actonel: Placebo Testosterone Patch and placebo Actonel tablet
Period: Overall Study
Arm/Group | Placebo Actonel and Active Testosterone Patch | Active Actonel and Active Testosterone Patch | Active Actonel and Placebo Testosterone | Placebo Testosterone Patch and Placebo Actonel
Started | 19 | 20 | 20 | 18
Completed | 17 | 16 | 15 | 11
Not Completed | 2 | 4 | 5 | 7
Not completed — Withdrawal by Subject | 1 | 4 | 5 | 6
Not completed — Physician Decision | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Actonel and Active Testosterone Patch | Active Actonel and Active Testosterone Patch | Active Actonel and Placebo Testosterone | Placebo Testosterone Patch and Placebo Actonel | Total
Number analyzed (Participants) | 19 | 20 | 20 | 18 | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 20 | 20 | 18 | 77
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.1 (7.3) | 25.2 (6.2) | 25.3 (6.3) | 26.9 (7.2) | 26.1 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 20 | 20 | 18 | 77
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 20 | 20 | 18 | 77

OUTCOME MEASURES:

1. Primary Outcome: Bone Mineral Density
Description: Percent change in postero-anterior (PA) spine bone mineral density as measured by dual energy x-ray absorptiometry (DXA)over a 12-month period. The differences in log-transformed values are reported as percent change.
Time Frame: Baseline and 12 months
Population: 1 subject was excluded from analysis. A factorial analysis was performed and determines the effect of each intervention separately, whether or not a subject received the 2nd intervention. Therefore, data from all 76 subjects who participated were used to determine the effect of each intervention on our endpoints.
Measure: Mean (95% Confidence Interval); unit: percent change
Groups:
- Actonel (Risedronate) 35 mg Weekly: Actonel (risedronate) 35 mg, 1 tablet weekly
- Testosterone: Testosterone, initial dose 150 mcg transdermal daily, increased to 300 mcg daily in women with free testosterone levels below the median (n=25 women)
Arm/Group | Actonel (Risedronate) 35 mg Weekly | Testosterone
Number analyzed (Participants) | 40 | 39
percent change | 3.2 [1.8 to 4.6] | -0.6 [-2.0 to 0.8]
Statistical Analysis 1: Comparison: Actonel (Risedronate) 35 mg Weekly; Factorial analysis; Test type: Superiority or Other; p < 0.0001, Factorial analysis — This p value was for the effect of Actonel (risedronate) on bone mineral density of the spine; Percent change between 0 and 12 months = 3.2, 95% CI 2-sided [1.8 to 4.6]
Statistical Analysis 2: Comparison: Testosterone; Factorial analysis; Test type: Superiority or Other; p = 0.41, Factorial analysis — This p value was for the effect of testosterone on bone mineral density of the spine; Percent change between 0 and 12 months = -0.6, 95% CI 2-sided [-2.0 to 0.8]

2. Secondary Outcome: Markers of Bone Metabolism
Description: type 1 collagen C-telopeptide(CTX); The differences in log-transformed values are reported as percent change.
Time Frame: Baseline to 12 months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: percent change of CTX
Groups:
- Actonel (Risedronate): Actonel (risedronate) 35 mg tablet weekly
- Testosterone: Testosterone patch(starting dose 150 mcg daily; increased to 300 mcg daily in subjects whose levels remained below the median on the initial dose)
Arm/Group | Actonel (Risedronate) | Testosterone
Number analyzed (Participants) | 40 | 39
percent change of CTX | -41 [-65 to -17] | -11 [-35 to 13]
Statistical Analysis 1: Comparison: Actonel (Risedronate); Factorial analysis; Test type: Superiority or Other; p = 0.002, Factorial analysis — This p value was for the effect of Actonel (risedronate); Percent change between 0 and 12 months = -41
Statistical Analysis 2: Comparison: Testosterone; Factorial analysis; Test type: Superiority or Other; p = 0.39, Factorial analysis — This p value was for the effect of testosterone; Percent change between 0 and 12 months = -11

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Placebo Actonel and Active Testosterone Patch | Active Actonel and Active Testosterone Patch | Active Actonel and Placebo Testosterone | Placebo Testosterone Patch and Placebo Actonel
Serious Adverse Events (participants affected / at risk) | 6/19 | 1/20 | 5/20 | 2/18
Other Adverse Events (participants affected / at risk) | 12/19 | 16/20 | 16/20 | 12/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Actonel and Active Testosterone Patch (N=19) | Active Actonel and Active Testosterone Patch (N=20) | Active Actonel and Placebo Testosterone (N=20) | Placebo Testosterone Patch and Placebo Actonel (N=18)
Hospitalization related to underlying condition (anorexia nervosa) (Psychiatric disorders) | 6 (16) | 1 (11) | 5 (13) | 2 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Actonel and Active Testosterone Patch (N=19) | Active Actonel and Active Testosterone Patch (N=20) | Active Actonel and Placebo Testosterone (N=20) | Placebo Testosterone Patch and Placebo Actonel (N=18)
Mild irritation at patch site (Skin and subcutaneous tissue disorders) | 9 (18) | 11 (27) | 8 (29) | 7 (15)
Mild increase in acne or oily skin (Skin and subcutaneous tissue disorders) | 8 (21) | 13 (28) | 13 (33) | 12 (33)
Mild increase in body hair growth (Skin and subcutaneous tissue disorders) | 6 (11) | 7 (12) | 3 (4) | 3 (14)
Myalgias (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (2) | 2 (2) | 0 (0)
Reflux (Gastrointestinal disorders) | 5 (8) | 3 (8) | 1 (3) | 6 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No